CLINICAL TRIAL: NCT03529669
Title: Evaluation of a Non-Endoscopic Immunocytological Device (Cytosponge™) for Post Chemo-radiotherapy Surveillance in Patients With Oesophageal Cancer -a Feasibility Study.
Brief Title: Cytosponge™ for Post-Chemoradiation Surveillance of Oesophageal Cancer
Acronym: CYTOFLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Centre for Statistics in Medicine (Other); Cancer Research UK (Other); University of Cambridge (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OCTO_068
Record Dates: First submitted 2018-02-26; First posted 2018-05-18 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-03

CONDITIONS: Oesophageal Cancer
Keywords: Cancer; Oesophageal Cancer; Gastrointestinal
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cytosponge™ (Experimental): All participants will receive the Cytosponge™ device.
  Interventions: Device: Cytosponge™

INTERVENTIONS:
Device: Cytosponge™ — Cytosponge™ is a capsule-sized device which contains an expandable, spherical mesh which is attached to a string. The capsule dissolves in the stomach after swallowing, releasing the sponge which is then retrieved by gently pulling the string after five minutes. As the sponge is pulled out it collects the cells from the lining of the gullet.

SUMMARY:
This is a feasibility study testing the use of the Cytosponge™ device in patients with known oesophageal cancer treated with pre-operative or definitive chemoradiation. All participants will receive one Cytosponge™ procedure at one time-point within 4-16 weeks after completion of chemoradiotherapy.

DETAILED DESCRIPTION:
In this feasibility study, we are investigating a novel way to test for remaining or reoccurring oesophageal cancer following chemoradiotherapy. The technique used to test this is called a Cytosponge™. We will be testing the use of the Cytosponge™ to determine completion rate, safety and acceptability of the procedure.

Cytosponge™ is a capsule-sized device which contains an expandable, spherical mesh which is attached to a string. The capsule dissolves in the stomach after swallowing, releasing the sponge which is then retrieved by gently pulling the string after five minutes. As the sponge is pulled out it collects the cells from the lining of the gullet.

The Cytosponge™ will be processed for evidence of residual cancer through analysis of cellular atypia and molecular biomarkers. Where available, the results will be compared with histology.

Up to fifty patients will be recruited to the trial across 11 sites.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age >/=16 years who

   1. have undergone pre-operative CRT as treatment for oesophageal cancer and due to undergo oesophagectomy or
   2. have undergone definitive CRT as treatment for oesophageal cancer
2. 4-16 weeks post completion of CRT
3. Dysphagia score 0-2 (Mellow Scale)*
4. Able to swallow tablets
5. Physiologically fit for endoscopy
6. Written (signed and dated) informed consent
7. The patient is willing and able to comply with the protocol for the duration of the study, and scheduled follow-up visits and examinations.

Exclusion Criteria:

1. Known to have oesophageal varices or stricture requiring dilatation of the oesophagus.
2. Unable to temporarily discontinue anticoagulation therapy/medication prior to their procedure*
3. Oesophageal stent
4. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor study candidate or could interfere with protocol compliance or the interpretation of study results.

   * Patients on anti-coagulation therapy are eligible for the study as long as they are considered suitable candidates for endoscopic biopsy (follow local hospital procedures for management of patients on anticoagulation due to undergo endoscopy). If temporary discontinuation of anticoagulation is required, this should be after consultation with the patients clinical care team.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Somnath Mukherjee, Principal Investigator — University of Oxford
Locations (11):
- United Kingdom (11):
  - Glan Clwyd hospital, Bodelwyddan
  - Cancer Institute Bristol, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Castle Hill hospital, Hull
  - Leicester General hospital, Leicester
  - The Christie, Manchester
  - Clatterbridge hospital, Metropolitan Borough of Wirral
  - Milton Keynes University Hospital, Milton Keynes
  - Churchill hospital, Oxford
  - University Hospital Southampton, Southampton

REFERENCES:
- [Derived] Jones CM, O'Connor H, O'Donovan M, Hayward D, Blasko A, Harman R, Malhotra S, Debiram-Beecham I, Alias B, Bailey A, Bateman A, Crosby TDL, Falk S, Gollins S, Hawkins MA, Kadri S, Levy S, Radhakrishna G, Roy R, Sripadam R, Fitzgerald RC, Mukherjee S. Use of a non-endoscopic immunocytological device (Cytosponge) for post chemoradiotherapy surveillance in patients with oesophageal cancer in the UK (CYTOFLOC): A multicentre feasibility study. EClinicalMedicine. 2022 Sep 23;53:101664. doi: 10.1016/j.eclinm.2022.101664. eCollection 2022 Nov. PMID 36187722

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytosponge™
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cytosponge™
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.32 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Dysphagia level [Count of Participants; unit: Participants]
  Able to eat normal diet / no dysphagia | 27
  Able to swallow some solid foods | 12
  Able to swallow only semi-solid foods | 2
Chemo-radiotherapy [Count of Participants; unit: Participants]
  Definitive chemo-radiotherapy | 28
  Neo-adjuvant chemo-radiotherapy | 13
Tumour site [Count of Participants; unit: Participants]
  Oesophagogastric junction | 4
  Lower thoracic oesophagus | 22
  Middle thoracic oesophagus | 8
  Upper thoracic oesophagus | 7
Tumour type [Count of Participants; unit: Participants]
  Adenocarcinoma | 16
  Squamous cell carcinoma | 25
WHO performance status [Count of Participants; unit: Participants]
  0 = Able to carry out normal activity without restriction | 26
  1 = Restricted in strenuous activity but ambulatory and able to carry out light work | 15

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate
Description: The percentage of consented, evaluable patients successfully undergoing the Cytosponge™ procedure.
Time Frame: Day 1 following intervention
Population: Individuals who attempted to carry out the Cytosponge procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cytosponge™
Number analyzed (Participants) | 41
Participants | 39

2. Secondary Outcome: Safety; Number of SAEs Related to the Device Procedure
Description: All serious adverse effects related to the procedure, including bleeding (requiring transfusion) and perforation.
Time Frame: Two week follow up
Population: The participants who successfully swallowed the Cytosponge device (i.e. 2 participants in the total population of 41 did not manage to do so).
Measure: Number; unit: events
Arm/Group | Cytosponge™
Number analyzed (Participants) | 39
events | 2

3. Secondary Outcome: Number of Participants With Positive Cytosponge™ Results From Biomarker Analysis (i.e. Presence of Cytological Atypia and/or p53 Abnormality)
Description: Quality of material obtained from Cytosponge™ test was centrally analysed at Cambridge (cellularity, yield and quality of extracted DNA as measure of quality). A positive Cytosponge™ result was defined as presence of positive cytological atypia, atypia of uncertain significance, and/or p53 aberrant.
Time Frame: From sample taken from Cytosponge™ on day of intervention
Population: Cytosponges suitable for biomarker analysis (i.e. 1 of the 39 swallowed devices was not analysed).
Measure: Count of Participants; unit: Participants
Arm/Group | Cytosponge™
Number analyzed (Participants) | 38
Participants | 9

4. Secondary Outcome: Acceptance Rate
Description: Percentage of eligible patients approached who consented.
Time Frame: Day 1 after questionnaire completion
Population: Of the 101 individuals who were initially identified as being eligible for CYTOFLOC, 96 were approached for consent to participate.
Measure: Count of Participants; unit: Participants
Arm/Group | Cytosponge™
Number analyzed (Participants) | 96
Participants | 41

5. Secondary Outcome: Number of Patients Who Would be Prepared to Repeat the Procedure
Description: Number of patients who have successfully undergone the procedure & would be prepared to accept the procedure repeatedly if it was to be used for follow-up (data captured through questionnaire after procedure).
Time Frame: Day 1 after questionnaire completion
Population: Participants who successfully completed the Cytosponge procedure (out of a total of 41 who attempted it).
Measure: Count of Participants; unit: Participants
Arm/Group | Cytosponge™
Number analyzed (Participants) | 39
Participants | 37

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Cytosponge administration to completion of the 2 week telephone follow up interview.
Description: The Cytosponge is an Investigational Medical Device & therefore additional categorisation of Adverse Device Effect (ADE) and Serious Adverse Device Effect (SADE) was required. Of the 41 trial participants, 39 successfully swallowed the Cytosponge device and were therefore evaluable for Adverse Events.
Arm/Group | Cytosponge™
All-Cause Mortality (participants affected / at risk) | 3/39
Serious Adverse Events (participants affected / at risk) | 1/39
Other Adverse Events (participants affected / at risk) | 3/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytosponge™ (N=39)
Acute cholecystitis (Hepatobiliary disorders) | 1 — Diagnosed 5 days after the Cytosponge procedure and persisting past the end of study. Defined as probably not related to the Cytosponge procedure.
Pneumonia (Infections and infestations) | 1 — Diagnosed 7 days after the Cytosponge procedure and persisting past the end of study. Defined as probably not related to the Cytosponge procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytosponge™ (N=39)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 — Starting on the day of Cytosponge procedure and persisting past the end of study. Classified as CTCAE grade 1 and probably not related to the procedure.
Dysphagia (Gastrointestinal disorders) | 1 — Starting 7 days following the Cytosponge procedure and resolving within 7 days. Classified as CTCAE grade 1 and probably not related to the procedure.
Dyspepsia (Gastrointestinal disorders) | 1 — Starting on the day of the Cytosponge procedure and resolving within 3 days. Classified as CTCAE grade 1 and possibly related to the procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
NHS Organisations shall not publish or otherwise disseminate the conclusions of the Study, including all or any part of the Results of the Study without prior written consent of the Sponsor, such consent not to be unreasonably withheld. Any publication or other dissemination of the conclusions of the Study by NHS Organisations shall not occur until the Sponsor has published the conclusions of the Study & shall refer to publication by the Sponsor in such form as the Sponsor may reasonably direct.

DOCUMENTS (2):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03529669/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03529669/SAP_001.pdf